CLINICAL TRIAL: NCT00957892
Title: Effects of Infant Formula Composition on Infant Feeding Behaviors
Status: Completed | Type: Observational
Sponsor: Monell Chemical Senses Center (Other)
Collaborators: Ajinomoto USA, INC. (Industry); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Julie A. Mennella, Member, Monell Chemical Senses Center
Other Study IDs: 809649; R01HD037119 (NIH); F32HD063343-01A1 (NIH)
Record Dates: First submitted 2009-08-12; First posted 2009-08-13 (Estimated); Last update posted 2017-12-18 (Actual); Status verified 2017-12

CONDITIONS: Healthy Infants
Keywords: Healthy Infants; Satiation; Satiety; Intake Regulation; Infant Feeding; Infant Formula Feeding

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — DNA collected for analysis of taste receptor and obesity-related genes
Oversight: Data Monitoring Committee: No

SUMMARY:
There is a paucity of information on whether and how the composition of formulas fed to infants influences their short-term feeding behaviors during the first few months of life. The purpose of this study is to investigate whether the composition of infant formula affects infants' feeding behaviors, in particular, how much formula is consumed within a given feed (i.e., measure of satiation) and how much time elapses after the feed until the infant exhibits signs of hunger (i.e., measure of satiety). The investigators will also examine the relationship between the composition of infant formula consumed and infant temperature, activity, sleep, and mothers' perceptions of infants' intake and regulatory behaviors.

DETAILED DESCRIPTION:
This is a within-subject, 3-day study. Each mother-infant dyad will visit the Monell Center three times, for 5 hours each time. The protocol during the three visits will be identical. Upon arrival, the infant will be changed into a light-weight cotton body suit. Infants and mothers will be weighed and measured for height. An activity sensor will be placed on the infant and temperature sensors will be placed on both the infant and the mother. When the infant signals hunger, he/she will be fed one of three formulas in randomized order:

1. cow milk based-formula (Enfamil)
2. protein hydrolysate formula (Nutramigen)
3. cow milk-based formula with glutamate level similar to Nutramigen (Enfamilg)

Intake will be monitored and all feeds will be videotaped. In between feedings, infants will rest or sleep on their backs in a crib and mothers will fill out questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, term infants of any racial background
* Infants may be of either sex
* Infants must be between 1 and 4 months of age
* Infants must be exclusively feeding a cow's milk-based formula
* Mothers must be over 18 years of age

Exclusion Criteria:

* Infants who were preterm
* Infants who have medical conditions that interfere with feeding or eating
* No major complications during pregnancy or at birth

Ages: 1 Month to 4 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Mothers with healthy infants who are between the ages of 1 to 4 months and are exclusively feeding cows milk-based formulas will be recruited from the Philadelphia area for this within-subject experimental research study.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2009-05; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Satiation: volume of formula consumed within a feed | 5-hour period
Satiety: the duration between feedings | 5-hour period

SECONDARY OUTCOMES:
Infant temperature change | 5-hour period
Infant sleep and activity patterns | 5-hour period
Maternal perceptions | 5-hour period

CONTACTS AND LOCATIONS:
Overall Officials: Julie A Mennella, Ph.D., Principal Investigator — Monell Chemical Senses Center
Locations (1):
- Monell Chemical Senses Center, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Mennella JA, Beauchamp GK. Developmental changes in the acceptance of protein hydrolysate formula. J Dev Behav Pediatr. 1996 Dec;17(6):386-91. doi: 10.1097/00004703-199612000-00003. PMID 8960567
- [Derived] Ventura AK, Beauchamp GK, Mennella JA. Infant regulation of intake: the effect of free glutamate content in infant formulas. Am J Clin Nutr. 2012 Apr;95(4):875-81. doi: 10.3945/ajcn.111.024919. Epub 2012 Feb 22. PMID 22357724